CLINICAL TRIAL: NCT05222178
Title: A Phase 1, Open-Label, Dose-Escalation Study to Evaluate the Safety and Efficacy of HMI-103 Administered Intravenously in Adult Participants With Classical PKU Due to PAH Deficiency
Brief Title: Safety and Efficacy of HMI-103 in Participants With Classical PKU Due to PAH Deficiency
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Homology Medicines Inc. has discontinued the development of this program.
Sponsor: Homology Medicines, Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HMI-103-101
Record Dates: First submitted 2021-12-21; First posted 2022-02-03 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Phenylketonurias; PAH Deficiency; Phenylketonuria
Keywords: PKU; Gene editing; AAVHSC
MeSH Terms: conditions — Phenylketonurias

STUDY DESIGN:
Intervention Model Description: Dose Escalation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Low Dose Cohort (Experimental): HMI-103 delivered IV one time
  Interventions: Drug: HMI-103
- Intermediate Dose Cohort (Experimental): HMI-103 delivered IV one time
  Interventions: Drug: HMI-103
- High Dose Cohort (Experimental): HMI-103 delivered IV one time
  Interventions: Drug: HMI-103

INTERVENTIONS:
Drug: HMI-103 — HMI-103 is an AAVHSC15 capsid containing a functional copy of the human PAH gene

SUMMARY:
This is an open-label, sequential ascending dose-escalation, Phase 1 study to evaluate the safety and efficacy of a single intravenous (I.V.) administration of HMI-103, a gene editing development candidate, in adult participants aged 18 to 55 years, inclusive, with classical PKU due to PAH deficiency who have uncontrolled disease despite Phe restricted dietary management.

DETAILED DESCRIPTION:
This is an open-label, sequential ascending dose-escalation, Phase 1 study to evaluate the safety and efficacy of a single intravenous administration of HMI-103, a gene editing development candidate, in adult participants aged 18 to 55 years, inclusive, with classical PKU due to PAH deficiency who have uncontrolled disease despite Phe-restricted dietary management. Up to 3 dose levels of HMI-103 may be investigated. At a given dose level, 3 participants are planned to be enrolled and dosed. Participant dosing will be staggered.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18-55 years of age at the time of informed consent
* Diagnosis of classical phenylketonuria (PKU) due to PAH deficiency
* Four baseline plasma Phe values with a concentration of ≥ 600 μmol/L and at least one historical value ≥ 600 μmol/L in the preceding 24 months.
* Participants must have uncontrolled classical PKU disease (despite Phe-restricted dietary management) in the judgment of the investigator and confirmed by the independent DMC at the end of the Screening period.
* Participant has the ability and willingness to maintain their baseline diet, for the duration of the trial, unless otherwise directed

Exclusion Criteria:

* Subjects with PKU that is not due to PAH deficiency
* Presence of anti-AAVHSC15 neutralizing antibodies
* Participants who are well controlled on a Phe-restricted diet.
* Hemoglobin A1c >6.5% or fasting glucose >126 mg/dL
* Liver function tests > ULN
* International normalized ratio (INR) > 1.2
* Hematology values outside of the normal range
* Previously received gene therapy for the treatment of any condition.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 3 (Actual)
Dates: Start 2022-06-03 (Actual); Primary Completion 2023-09-14 (Actual); Study Completion 2023-09-14 (Actual)

PRIMARY OUTCOMES:
To measure incidence and severity of Treatment Emergent Adverse Events (TEAEs) and adverse events of special interest (AESIs) of a single administration of HMI-103 | Baseline to Week 104
To evaluate the efficacy of HMI-103 on reduction of plasma Phe concentration at each dose level | Baseline to Weeks 24-32
  Mean percent change from baseline at Weeks 24-32 in plasma Phe concentration within each dose cohort post-administration of HMI-103

SECONDARY OUTCOMES:
To evaluate the effect of HMI-103 on plasma Phe concentration relative to treatment guidelines for PKU | Baseline to Week 104
  Incidence of plasma Phe of ≤ 360 μmol/L within each dose cohort at each timepoint post-administration of HMI-103
To assess durability of response | Weeks 48-52
  Incidence of plasma Phe ≤ 360 μmol/L during Weeks 48-52 post-administration of HMI-103
To assess the changes in dietary protein intake | Baseline to Week 104
  Change from baseline in natural and total protein intake (g/day) at each timepoint post-administration of HMI-103

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - The Community Health Clinic, Topeka, Indiana
  - Clinic for Special Children, Lancaster, Pennsylvania